CLINICAL TRIAL: NCT03091062
Title: Evaluation of the Effectiveness of the Monarch™ Airway Clearance System as Determined by Mucus Production
Brief Title: Evaluation of an Airway Clearance System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLUI-2016-182
Record Dates: First submitted 2017-02-14; First posted 2017-03-27 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Group (Experimental): Study subjects will serve as their own control and all will receive treatment with two different Airway Clearance Systems- the Vest® Airway Clearance System and the Monarch™ System. Subjects will be randomized to which treatment is received first.
  Interventions: Device: Vest® Airway Clearance System; Device: Monarch™ System

INTERVENTIONS:
Device: Vest® Airway Clearance System — High frequency chest wall oscillation (HFCWO) therapy is commonly prescribed to provide routine airway clearance in patients with a need for regular airway clearance therapy. HFCWO generates high velocity expiratory airflow that is thought to mobilize secretions by the sheer force created.
Device: Monarch™ System — Generates airflow at frequencies similar to those provided by HFCWO and also provides direct percussive therapy.

SUMMARY:
The aim of this study is to assess the effectiveness of an Airway Clearance System.

DETAILED DESCRIPTION:
The study will compare the effectiveness of The Monarch™ System and The Vest® Airway Clearance System. All subjects will receive treatment with both systems and endpoints will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Cystic Fibrosis (CF) (by sweat test and/or genetics)
* Age ≥ 15 years
* Ability to expectorate sputum daily - determined by treating physician
* Patient must be on a stable regimen of CF medication for 4 weeks prior to Visit 1
* Patient who requires regular home airway clearance therapy

Exclusion Criteria:

* Forced Expiratory Volume in 1 Second (FEV1) < 30 % predicted or > 90 % predicted
* Anticipated requirement for hospitalization within the next three weeks
* History of pneumothorax within the past 6 months prior Visit 1
* History of haemoptysis requiring embolization within the past 12 months prior to Visit 1
* Inability to perform Monarch™ and/or Vest® System therapy as directed
* Unable or unwilling to complete study visits or provide follow-up data as required per the study protocol
* Has taken Intravenous (IV) antibiotics within the past 4 weeks prior to Visit 1
* Has ongoing exacerbation or Allergic bronchopulmonary aspergillosis (ABPA)
* Pregnant or lactating female
* Has a pacemaker or implantable cardioverter defribillator (ICD)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Wet Weight of Sputum Produced | Through study completion, an average of 2 months
  Assessment of the wet weight of total sputum that is produced as a result of each of two therapy sessions. The total wet weight includes the wet weight of sputum collected each 30-minute therapy session + the wet weight of sputum collected during a 1-hour collection period following each therapy.

SECONDARY OUTCOMES:
Sputum Volume | Through study completion, an average of 2 months
  Assessment of the total volume of sputum that is produced as a result of each of two therapy sessions. The total volume includes the volume of sputum collected each 30-minute therapy session + the volume of sputum collected during a 1-hour collection period following each therapy.
Functional Respiratory Imaging | Through study completion, an average of 2 months
  Functional Respiratory Imaging will be completed utilizing CT scans. The CT scans are to be completed before airway clearance therapy on each day and after the one-hour sputum collection following the airway clearance therapy (a minimum of one hour following completion of the airway clearance therapy).
Brody Scores (Scoring of CT Scans) | Through study completion, an average of 2 months
  Brody Scores will be completed utilizing CT scans. The CT scans are to be completed before airway clearance therapy on each day and after the one-hour sputum collection following the airway clearance therapy (a minimum of one hour following completion of the airway clearance therapy).
Lung Clearance Index | Through study completion, an average of 2 months
  Measurement of how much ventilation is required to completely clear the full residual capacity using the Inert Gas Multi-Breath Washout method completed pre- and post-therapy -- before the airway clearance therapy on each day and after the one-hour sputum collection following the airway clearance therapy (a minimum of one hour following completion of the airway clearance therapy).
Subjective satisfaction surveys | Through study completion, an average of 2 months
  Patient satisfaction with therapy will be assessed post therapy. (survey will be completed a minimum of one hour following completion of the airway clearance therapy).
Spirometry | Through study completion, an average of 2 months
  Forced expiratory spirometry maneuvers will be completed before and after therapy. -- before the airway clearance therapy on each day and after the one-hour sputum collection following the airway clearance therapy (a minimum of one hour following completion of the airway clearance therapy).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No